CLINICAL TRIAL: NCT02322268
Title: Metabolomic Profiling on The Effect of Cosmos Caudatus (Ulam Raja) Supplementation in Patients With Type 2 Diabetes: A Randomized Controlled Trial
Brief Title: RCT Evaluating Effects of Cosmos Caudatus (Ulam Raja) in T2DM Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Cheng Shi Hui, Cheng Shi Hui, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6370700
Record Dates: First submitted 2014-12-20; First posted 2014-12-23 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Type 2 Diabetes Mellitus; Obesity
Keywords: Type 2 Diabetes Mellitus; Cosmos Caudatus; Ulam Raja; Metabolomic profiling; antioxidant
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Diabetic Cosmos caudatus treated group (Experimental): Subjects in this arm will receive Cosmos caudatus for 8 weeks.
  Interventions: Dietary Supplement: Cosmos Caudatus
- Diabetic control group (No Intervention): Subject in this group will not receive Cosmos caudatus. However, they will be educated for the same calorie intake and lifestyle intervention as in Cosmos caudatus treated group.

INTERVENTIONS:
Dietary Supplement: Cosmos Caudatus — 15g of Cosmos caudatus consumed with lunch or dinner
  Other Names: Ulam Raja
  Arms: Diabetic Cosmos caudatus treated group

SUMMARY:
The purpose of this study is to determine whether Cosmos caudatus is effective as an adjuvant therapy for type 2 Diabetes Mellitus.

DETAILED DESCRIPTION:
Background: Cosmos caudatus (C. caudatus) ethanol extract has been reported to have extraordinary high antioxidant capacity compared to other plants. Furthermore it has been shown to reduce the plasma blood glucose and lipid profile significantly in an animal model. However, no study has been reported on its effectiveness in human. Therefore, we plan to conduct a randomized controlled trial to evaluate the effectiveness and safety of C. caudatus on glycemic status, oxidative stress markers, inflammatory markers, lipid profile in patients with type 2 diabetes. Besides, metabolomics approach will be carried out to compare the metabolite changes between diabetic C. caudatus treated and control patients.

Methods: A single-center randomized, controlled, two-arm parallel design clinical trial will be carried out in Malaysia. This study enrol 92 patients diagnosed with type 2 diabetes. Diabetic patients who meet eligibility criteria will be randomly allocated to two groups, which are C. caudatus treatment group and control group. Both groups will be compared on the primary and secondary outcomes at baseline, 4, 8, and 12 weeks. The serum and urine metabolome of both groups will be examined using proton NMR spectroscopy.

Discussion: The study will provide insights into the potential beneficial effect of C. caudatus in type 2 diabetic patients. In addition, the therapeutic effect of C. caudatus towards type 2 diabetes will reflect as a change of metabolite profile in urine and serum.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed type 2 diabetes with at least 6 months diagnosis
2. BMI between 18.5-40 kg/ m2
3. Able to comply to the study protocol
4. They are treated with stabilized dose of oral diabetic agents

Exclusion Criteria:

1. Pregnant and lactating
2. Have any gastrointestinal disorder that interferes the bowel function, severe hepatic or renal disease (dialysis), an infection that requires antibiotics within three weeks
3. They are currently on insulin regimen.
4. Individuals on the following drugs which will possibly have herb-drug interaction: anticoagulant such as warfarin and aspirin, corticosteroids (Prednisolone), fluoroquinolones (ciprofloxacin, levofloxacin), doxorubicin, cisplatin, cyclosporine, and digoxin

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2014-08; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Glycemic control | 1 month

SECONDARY OUTCOMES:
Liver profile | 1 month
Renal profile | 1 month
Blood pressure | 1 month
Metabolite profile | 1 month
Inflammatory marker | 1 month
Lipid profile | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Shi Hui Cheng, Principal Investigator — Universiti Putra Malaysia
Locations (1):
- Hospital Serdang, Serdang, Selangor, Malaysia

REFERENCES:
- [Derived] Cheng SH, Ismail A, Anthony J, Ng OC, Hamid AA, Yusof BN. Effect of Cosmos caudatus (Ulam raja) supplementation in patients with type 2 diabetes: Study protocol for a randomized controlled trial. BMC Complement Altern Med. 2016 Feb 27;16:84. doi: 10.1186/s12906-016-1047-7. PMID 26920910
- See also: Type 2 Diabetes — http://www.nlm.nih.gov/medlineplus/diabetestype2.html
- See also: Medlineplus — http://www.nlm.nih.gov/medlineplus/